CLINICAL TRIAL: NCT06085443
Title: Clinical Study to Evaluate the Safety and Effectiveness of an Auricular Spray Medical Device Ear Hygiene
Brief Title: Safety and Effectiveness of an Auricular Spray
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: YSLab (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23E1670
Record Dates: First submitted 2023-10-03; First posted 2023-10-17 (Actual); Results first posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Excessive Ear Wax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular spray (Experimental): Subjects using the medical device under investigation: 2 sprays in each ear, every 3 days at home.
  Interventions: Other: Ear Hygiene
- Control (No Intervention): Subjects not using any spray (can use ear drops in case of discomfort or pain)

INTERVENTIONS:
Other: Ear Hygiene — 2 sprays in each ear, every 3 days at home
  Arms: Auricular spray

SUMMARY:
The goal of this clinical trial is to test the safety and efficacy of a medical device in subjects with cerumen in excess. The main questions it aims to answer are:

* Does the medical device induce skin irritation in the ear canal?
* Does the medical device reduce obstruction of ear canal induced by excessive cerumen?

Participants will use the device in each ear, once a day, every 3 days at home. Researchers will compare the medical device group to a control group who will not use the medical device.

DETAILED DESCRIPTION:
Ocean Bio Actif Hygiène de l'oreille is a medical device class IIa indicated for the prevention of the formation of earwax plugs and consequently the pathologies linked to the accumulation of earwax (hearing loss and infection/affection of the external auditory canal).

This clinical investigation is designed to improve the quality and quantity of data available on both the safety and the efficacy of Ocean Bio-Actif, in order to confirm the safety and the efficacy of the product in a post-market environment.

The objective of the current clinical investigation is to confirm the efficacy and safety of topical application to the ear canal of Ocean Bio-Actif.

ELIGIBILITY:
Inclusion Criteria:

* Gender: female and/or male.
* Age:

  30 to 40% having age between 3 to 12 yo, 30 to 40% between 13 to 65 yo, 30 to 40% more than 65 yo.
* Subjects able to use the tested product.
* Subjects having history of cerumen occlusion more than once a year with or without symptoms (reduction of hearing function, obstruction feeling of the ear canal,..).
* Subjects having ear help system or regular users of systems such as anti-noise plugs or headsets (only for the 13yo subjects and more).
* Subjects having a clinical score of ear canal obstruction of 2 or 3 at D0.

Exclusion Criteria:

* Subjects who had chirurgical act on the mastoïde.
* Subjects who had severe troubles of the internal ear (severe dizziness, desorientation, nausea).
* Subjects using regularly a ear spray for washing his/her ears.
* Subjects having a score of ear canal obstruction at 4 at D0.
* Pregnant or nursing woman or planning a pregnancy during the study;
* Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship;
* Subject in a social or sanitary establishment;
* Subject suspected to be non-compliant according to the investigator's judgment;
* Subject with a condition or receiving a medication which, in the investigator's judgment, put the subject at undue risk;
* Subject suffering from a severe or progressive disease.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iwona MAZUREWICZ, Principal Investigator — Eurofins Dermscan
Locations (1):
- Eurofins Dermscan Poland, Gdansk, Ul. Matuszewskiego 12, Poland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment at the investigational sites
Pre-assignment Details: Each subject having signed a consent form will be assigned a "screening subject number" according to his/her chronological order of arrival in the study.
Period: Overall Study
Arm/Group | Auricular Spray | Control
Started | 64 | 35
Completed | 63 | 35
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: The overall Number of Baseline Participants does not differ from the number of participants assigned to the arm or comparison group and in the entire study population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Auricular Spray | Control | Total
Number analyzed (Participants) | 64 | 35 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 15 | 40
  Between 18 and 65 years | 23 | 11 | 34
  >=65 years | 16 | 9 | 25
Age, Continuous [Mean (Full Range); unit: years] | 36.2 [3 to 83] | 35.6 [3 to 76] | 36.2 [3 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 22 | 64
  Male | 22 | 13 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 64 | 35 | 99
Region of Enrollment [Number; unit: participants]
  Poland | 64 | 35 | 99

OUTCOME MEASURES:

1. Primary Outcome: Skin Irritation
Description: To confirm the safety of the device by clinical examination by ENT specialist and scoring of the irritation of the ear canal at Day90 in comparison with basal scoring of irritation at Day0 such as:
  * 0: no irritation,
  * 1: slight irritation (located slight erythema and/or dryness),
  * 2: moderate irritation (clear erythema or dryness which may be visible on the whole treated area),
  * 3: severe irritation (serious erythema with potential oedema and/or scar).
Time Frame: Day0 and Day90
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Auricular Spray | Control
Number analyzed (Participants) | 64 | 35
score on a scale
  Irritation at D0 | 0.22 (0.45) | 0.20 (0.41)
  Irritation D90 | 0.13 (0.49) | 0.11 (0.32)

2. Secondary Outcome: Ear Canal Obstruction Due to Excessive Earwax
Description: To confirm the efficacy/performance of the device for the prevention of ear obstruction in comparison to baseline (Day0) and between groups using the scoring of the obstruction of ear canal by the Investigator:
  0: no obstruction - normal and/or no significant presence of cerumen in the ear canal. The membrane is clearly visible.
  1. <25% minimal, very little and mostly insignificant impacted cerumen. The tympanic membrane is visible, but with still a little bit cerumen.
  2. 25-50% mild, some excessive impacted cerumen causing partial occlusion of the ear canal. The tympanic membrane is not entirely visible, quite difficult to see.
  3. 50-75% moderate, moderate and excessive impacted cerumen causing partial occlusion of the ear canal. Partial to very little of the tympanic membrane is visible.
  4. 75-100% severe, severe and excessive impacted cerumen causing partial or complete occlusion of the ear canal. Little if any of the tympanic membrane is visible.
Time Frame: Day0 and Day90
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Auricular Spray | Control
Number analyzed (Participants) | 63 | 35
score on a scale
  Obstruction at D0 | 2.33 (0.48) | 2.29 (0.46)
  Obstruction at D90 | 1.19 (1.16) | 1.97 (0.92)

3. Secondary Outcome: Hearing Function
Description: Secondary aims: EFFICACY/PERFORMANCE PREVENTION for investigational device and for control group, in comparison to the baseline (Day0) using an audiogram (only for subjects more than 6).
  Hearing function was assessed in patients on day 0 (D0) and day 90 (D90). The mean difference in hearing function (D90 - D0), expressed in decibels (dB), was reported in a data table. A mean difference greater than +5 dB is considered a gain in hearing function, while a mean difference less than -5 dB is considered a loss in hearing function. A difference in hearing function within the range [-5 dB; +5 dB] is considered to indicate no effect on hearing function.
Time Frame: Day0 and Day90
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Auricular Spray | Control
Number analyzed (Participants) | 63 | 35
dB | 1.07 (5.69) | 0.26 (4.37)

ADVERSE EVENTS:
Time Frame: 90 days
Description: No serious adverse event is expected. No risk for mortality is expected.
Arm/Group | Auricular Spray | Control
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/35
Other Adverse Events (participants affected / at risk) | 1/64 | 0/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Auricular Spray (N=64) | Control (N=35)
itching (Ear and labyrinth disorders) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-09): https://cdn.clinicaltrials.gov/large-docs/43/NCT06085443/Prot_SAP_000.pdf